CLINICAL TRIAL: NCT04525300
Title: Changes of Gut Microbiome Following Liraglutide Treatment in Non-diabetic Obese Subjects or Overweight Subjects With Co-morbidities: A Randomised, Double-blind, Placebo Controlled, Parallel Group, Multi-centre, 28-week Trial
Brief Title: Gut Microbiome Changes Following Liraglutide Treatment in Obese Subjects or Overweight Subjects With Co-morbidities
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Wujing, professor, Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202005062
Record Dates: First submitted 2020-07-23; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Experimental): Subject receiving liraglutide 3.0 mg subcutaneous (under the skin) injection once daily for 28 weeks.
  Interventions: Drug: Liraglutide
- placebo (Placebo Comparator): Subject receiving placebo 3.0 mg subcutaneous (under the skin) injection once daily for 28 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Liraglutide — Randomization was performed with the use of a computer-generated system provided by the sponsor. Eligible patients were randomly assigned, in a 2:1 ratio, to receive once-daily subcutaneous injections of liraglutide, starting at a dose of 0.6 mg with weekly 0.6-mg increments to 3.0 mg, or placebo; both groups received counseling on lifestyle modification
  Other Names: S20200402
  Arms: Liraglutide
Drug: placebo — Randomization was performed with the use of a computer-generated system provided by the sponsor. Eligible patients were randomly assigned, in a 2:1 ratio, to receive once-daily subcutaneous injections of liraglutide, starting at a dose of 0.6 mg with weekly 0.6-mg increments to 3.0 mg, or placebo; both groups received counseling on lifestyle modification
  Other Names: S20200301
  Arms: placebo

SUMMARY:
We performed a multicenter, randomized, double-blind, placebo-controlled 28-week trial. 300 non-diabetic obese subjects or overweight subjects with co-morbidities were randomly assigned. Eligible participants were randomized 2:1 to once-daily subcutaneous injections of either liraglutide or placebo. The primary outcome is to investigate the composition of the gut microbiota from baseline to end of treatment.

DETAILED DESCRIPTION:
We performed a multicenter, randomized, double-blind, placebo-controlled 28-week trial. 300 individuals (18-75 years of age, body-mass index ≥30 kg/m2 or BMI 27-30kg/m2 accompanied by at least one weight-related complication (treated or untreated hypertension, dyslipidemia, pre-diabetes)) were randomly assigned. All the patients provided written informed consent before participation. Key exclusion criteria were type 1 or 2 diabetes, the use of medications that cause clinically significant weight gain or loss, previous bariatric surgery, a history of pancreatitis, a history of major depressive or other severe psychiatric disorders, and a family or personal history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma. Eligible participants were randomized 2:1 to once-daily subcutaneous injections of either liraglutide or placebo using a computer-generated, centrally administered procedure. Patients, investigators, and the sponsor were unaware of the study-group assignments. The primary outcome is to investigate the composition of the gut microbiota from baseline to end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activity takes place
* Obesity (BMI ≥30.0 kg/m2); or overweight (BMI ≥27.0 kg/m2) with treated or untreated co-morbid dyslipidemia (Low-density lipoprotein ≥3.38mmol/l (130 mg/dl), or triglycerides ≥1.7mmol/l (150 mg/dl), or high-density lipoprotein <1.04mmol/l (40 mg/dl) for males and <1.30mmol/l (50 mg/dl) for females) and/or hypertension (Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
* Age ≥18 years, ≤75 years

Exclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes per the judgment of the investigator
* HbA1c ≥6.5% or fasting plasma glucose ≥7.0 mmol/l or 2-hour post-challenge plasma glucose ≥11.1 mmol/liter (at screening)
* less than 5 kg self-reported change during the previous 3 months
* Previous treatment with GLP-1 receptor agonists (including liraglutide or exenatide) within the last 3 months
* Known or suspected hypersensitivity to trial product, related products or other GLP-1 receptor agonist
* Diet attempts using herbal supplements or over-the-counter medications within 1 months before screening, or use prescription drugs for weight loss within 3 months before screening (for example: orlistat, fenfluramine, maindole ) Or lipid dissolving injection (for example: lipolysis needle) treatment
* Current or history of treatment with medications that may cause significant weight gain, within 3 months prior to screening, including systemic corticosteroids (more than 1 week),tri-cyclic antidepressants, atypical antipsychotic and mood stabilizers (e.g. imipramine, amitriptiline, mirtazapin, paroxetine, phenelzine, clorpromazine, thioridazine, clozapine, lanzapine, valproic acid and its derivatives, and lithium)
* A history of malignant tumors within 5 years before screening (except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and ductal carcinoma in situ after radical operation)
* A history of severe heart disease is defined as: decompensated heart insufficiency (NYHA III-IV), and/or a history of unstable angina within 6 months before screening, and a history of myocardial infarction within 12 months
* Obesity induced by other endocrinologic disorders (e.g. Cushing's Syndrome)
* Suffer from gastrointestinal motility disorders or obstruction diseases, such as gastroparesis, gastroesophageal reflux disease
* Any lifetime history of a suicidal attempt or A history of any suicidal behavior in the last month prior to randomization
* A patient health questionnaire (PHQ-9) score of ≥15
* Montreal Cognitive Assessment Scale (MoCA) score <26 at screening;
* Any suicidal ideation of type 4 or 5 on the Columbian Suicidality Severity Rating Scale (C-SSRS) in the last month prior to randomization
* Untreated or uncontrolled hypothyroidism/hyperthyroidism defined as thyroid-stimulating hormone >6 mIU/liter or <0.4 mIU/liter
* Screening calcitonin ≥50 ng/liter
* Family or personal history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma (FMTC) or Personal history of non-familial medullary thyroid carcinoma
* History of chronic pancreatitis or idiopathic acute pancreatitis or amylase ≥ 3 times the upper limit of normal value during screening
* ALT or AST or TBiL>3 times the upper limit of normal value during screening
* Impaired renal function, defined as serum creatinine level ≥1.5mg/dL (132µmol/L) in men or ≥1.4mg/dL (123µmol/L) in women at screening
* Untreated or uncontrolled severe dyslipidemia, defined as blood LDL-C≥190mg/dl (4.94mmol/L) and/or TG≥500mg/dl (5.65mmol/L) at screening
* Uncontrolled treated/untreated hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg)
* Previous surgical treatment for obesity (excluding liposuction if performed >1 year before trial entry)
* According to the investigator's judgment, those who have a surgical plan during the trial period (except for minor operations)
* Participated in any weight loss clinical trials within 3 months before screening, and took any experimental drugs within 1 month (Re-screening is allowed once within the limit of the recruitment period)
* Known or suspected abuse of alcohol or narcotics within 6 months
* Poor compliance with restrictions on diet and behavior during screening
* Females of child-bearing potential who are pregnant, breast-feeding
* Participants intend to become pregnant or are not using adequate contraceptive methods or subjects who use hormonal contraceptives
* The investigator considers that it is not suitable for participants (for example, the investigator judges that severe obstructive sleep apnea will cause gastroesophageal reflux).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-05-24 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The composition of the gut microbiota from baseline to end of treatment. | week 28
  The composition of the gut microbiota from baseline to end of treatment compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China